CLINICAL TRIAL: NCT00810615
Title: Treatment of Moderate to Mild Cognitive Dysfunction Caused by Traumatic Brain Injury (TBI) With Hyperbaric Oxygen Therapy (HBOT)
Brief Title: Treatment of Traumatic Brain Injury With Hyperbaric Oxygen Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: San Antonio Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, George Wolf, Study Director, San Antonio Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FWH20080137H
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Results first posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2017-11

CONDITIONS: Brain Injury, Chronic
Keywords: chronic TBI; cognitive function; PTSD; HBO; hyperbaric; oxygen; chronic brain injury
MeSH Terms: conditions — Brain Injury, Chronic; Stress Disorders, Post-Traumatic | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham treatment (Sham Comparator): Subject will breathe air at less than 1.3 Atmospheres Absolute (ATA) in three 30 minute periods separated by 10 minutes of breathing air at less that 1.3 ATA. Hyperbaric exposures will be done up to 5 times per week with a total number of 30 exposures.
  Interventions: Other: Sham treatment
- Hyperbaric oxygen 2.4 ATA (Experimental): Subject will breathe 100% oxygen at 2.4 Atmospheres Absolute (ATA) in three 30 minute periods separated by 10 minutes of breathing air at 2.4 ATA. Hyperbaric exposures will be done up to 5 times per week with a total number of 30 exposures.
  Interventions: Other: Hyperbaric oxygen @ 2.4 ATA

INTERVENTIONS:
Other: Hyperbaric oxygen @ 2.4 ATA — Subject will breath 100% oxygen at 2.4 Atmospheres Absolute (ATA) in three 30 minute periods separated by 10 minutes of breathing air at 2.4 ATA. Hyperbaric exposures will be done up to 5 times per week with a total number of 30 exposures.
  Other Names: hyperbaric oxygen; HBOT; HBO
  Arms: Hyperbaric oxygen 2.4 ATA
Other: Sham treatment
  Other Names: sham exposure; 1.3 ATA air
  Arms: Sham treatment

SUMMARY:
The purpose of this study is to determine if hyperbaric oxygen therapy (HBOT) improves the cognitive function of OIF/OEF individuals who have chronic mild to moderate traumatic brain injury (TBI). Cognitive function includes such things as thinking, remembering, recognition, concentration ability and perception. Traumatic brain injury is common with head injuries caused by blows to the head, nearby explosions, or concussion. Subjects will be assigned to an intervention or sham arm. Computer based cognitive tests will be used as outcome measures. Subjects are enrolled by invitation only.

DETAILED DESCRIPTION:
The Agency for Healthcare Research and Quality (AHRQ) did a comprehensive review of the literature focusing on TBI, stroke and cerebral palsy in Sep 2003. The study design and goals were based on the AHRQ recommendations for future hyperbaric oxygen for TBI research. This report stated, "The most important gap in the evidence is a lack of a good quality time-series study or controlled trial of the effects of HBOT on cognition, memory, and functional status in patients with deficits due to mild and moderate chronic TBI." The AHRQ Evidence Report further stated, "Lack of agreement on the dosage of HBOT and the duration of treatment is an important barrier to conducting good-quality clinical studies…Good-quality dose-ranging studies of HBOT for brain injury can be done, based on the model used by pharmaceutical manufacturers and the FDA. It is likely that the dosage of HBOT needs to be individualized based on the patient's age, clinical condition, and other factors". Although there are many anecdotal cases of TBI improvement with HBO, this case is backed with non-subjective data. The biological basis for why breathing 100% oxygen under pressurized conditions improves chronic neurological trauma remains unclear. There is some evidence that chronic TBI effects are related to the demyelization effect linked to the expression of a specific protease, calpain. This protease is also seen in demyelination delayed effects of carbon monoxide poisoning which is slowed by treatment with HBO. The "idling neuron" theory advocated in neurological studies suggest that HBO may increase metabolic performance of chronically impaired neurons that were marginally capable, enabling restoration of full function leading in turn to increased integrative plasticity. HBO has been shown to increase recruitment of stem cells from the bone marrow, suggesting that HBO may increase the rate at which damaged neuronal tissue can be reconstituted de novo. The proposed research will treat 25 subjects using HBO (2.4 ATA breathing 100% oxygen) and 25 subjects in a sham HBO treatment (1.3 ATA breathing air). Computer-based cognitive testing and the Post-traumatic Stress Disorder Checklist for Military (PCL-M) will be administered pre- and post-HBOT as well as at intervals throughout the treatment. The cognitive test results and stem cell results will be analyzed within each subject at the various treatment points as well as cohort groups between each treatment leg. Cognitive test scores will also be compared to cognitive test population reference bases matched for gender and age. The Agency for Healthcare Research and Quality 2003 report also stated, "If there is a 1 percent chance that the treatment works, a rational decision maker would try it-there is a potential gain and no potential loss. On the other hand, if there are proven harms, and their severity and frequency are well described, the probability that the treatment works would have to be higher before most people would try it"

ELIGIBILITY:
Inclusion Criteria:

* neurology diagnosis of mild to moderate TBI
* injury sustained during OIF/OEF military activities
* perception of cognitive dysfunction following their injury
* stable mental status for at least two months
* stable psychotropic medication history for at least one month
* ability to perform computer based cognitive testing (must be capable using a mouse and PDA pointer and readily view the displays)
* TBI occurrence since 7 October 2001
* ability to consent

Exclusion Criteria:

* medical conditions that prevent subject from participating in hyperbaric environments
* previous hyperbaric oxygen treatments since being diagnosed with TBI
* history of alcohol abuse
* history of drug abuse

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. George Wolf, M.D., Study Director — SAMMC Hyperbaric Medicine; Leonardo C Profenna, M.D., Principal Investigator — SAMMC Hyperbaric Medicine

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from Nov 2008 - Nov 2010. Candidate subjects with a diagnosis of chronic truamatic brain injury (TBI) were identified by DoD neurologists. Those interested were screened for inclusion/exclusion criteria. 103 candidates were screened. 22 did not qualify; 31 were deferred (psychotropic medication or mental status unstable).
Groups:
- Sham Treatment: Subjects breathed air at less than 1.3 Atmospheres Absolute (ATA) in three 30 minute periods separated by 10 minutes of breathing air at less that 1.3 ATA. Hyperbaric exposures were done up to 5 times per week with a total number of 30 exposures. Pressurization time was seven minutes to a depth of 11 feet of sea water (fsw) or 1.3 ATA. The chamber pressure was slowly decreased over 10 minutes to 6 fsw (1.2 ATA). The final depressurization to surface was done over a 10 minute period. To simulate the treatment 2.4 ATA pressurization, pressurizations and depressurizations were done using venting techniques that would be nearly identical with the noise and temperature as that experienced with the treatment pressure. The inside observers simulated pressure equalization measures (Valsalva) every 10 to 30 seconds and breathed oxygen by mask (required in the 2.4 ATA pressure to prevent decompression sickness) at the same frequency as if they were in the treatment exposure pressure.
- Hyperbaric Oxygen 2.4 ATA: Subject breathed 100% oxygen at 2.4 Atmospheres Absolute (ATA) in three 30 minute periods separated by 10 minutes of breathing air at 2.4 ATA. Hyperbaric exposures were done up to 5 times per week with a total number of 30 exposures. Pressurization time was seven minutes to a depth of 45 feet of sea water (fsw) or 2.4 ATA. The final depressurization to surface was done over a 10 minute period. Inside observers used pressure equalization measures (Valsalva) every 10 to 30 seconds and breathed oxygen by mask (required in the 2.4 ATA pressure to prevent decompression sickness) three times (10/15/5 minute durations) during the exposure.
Period: Overall Study
Arm/Group | Sham Treatment | Hyperbaric Oxygen 2.4 ATA
Started | 25 | 25
Completed | 24 (One male withdrawal due to personal reasons.) | 24 (One male withdrawal due to personal reasons.)
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Sham Treatment: Subjects breathed air at less than 1.3 Atmospheres Absolute (ATA) in three 30 minute periods separated by 10 minutes of breathing air at less that 1.3 ATA. Hyperbaric exposures were done up to 5 times per week with a total number of 30 exposures. Pressurization time was seven minutes to a depth of 11 feet of sea water (fsw) or 1.3 ATA. The chamber pressure was slowly decreased over 10 minutes to 6 fsw (1.2 ATA). The final depressurization to surface was done over a 10 minute period. To simulate the treatment 2.4 ATA pressurization, pressurizations and depressurizations were done using venting techniques that would be nearly identical with the noise and temperature as that experienced with the treatment leg. The inside observers simulated pressure equalization measures (Valsalva) every 10 to 30 seconds and breathed oxygen by mask (required in the 2.4 ATA pressure to prevent decompression sickness)at the same frequency as if they were in the treatment exposure pressure.
- Hyperbaric Oxygen 2.4 ATA: Subject breathed 100% oxygen at 2.4 Atmospheres Absolute (ATA) in three 30 minute periods separated by 10 minutes of breathing air at 2.4 ATA. Hyperbaric exposures were done up to 5 times per week with a total number of 30 exposures. Pressurization time was seven minutes to a depth of 45 feet of sea water (fsw) or 2.4 ATA. The final depressurization to surface was done over a 10 minute period. Inside observers used pressure equalization measures (Valsalva) every 10 to 30 seconds and breathed oxygen by mask (required in the 2.4 ATA pressure to prevent decompression sickness) three times (10/15/5 minute durations)during the exposure.
- Total: Total of all reporting groups
Arm/Group | Sham Treatment | Hyperbaric Oxygen 2.4 ATA | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.4 (7.4) | 28.3 (8.1) | 28.3 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 24 | 24 | 48
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Computer Cognitive Test Scores - ImPACT Verbal Memory
Description: The Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT) battery was developed at the University of Pittsburgh. It has a sensitivity of 81.9% and specificity of 89.4% in discriminating between concussion and non-concussion groups. It consists of a medical history questionnaire regarding concussions and resultant symptoms including loss of consciousness, memory loss, confusion, headache, seizure activity, emotional state, and sleep patterns. There are four subtests given and scored by computer. These include verbal and visual memory, visual motor speed, and response time. The composite scores are specifically designed to determine changes within the individual, better or worse, over time. The verbal memory score demonstrates improvement as the score increases. The score range was 36.8 to 98.6.
Time Frame: Baseline and six weeks post hyperbaric exposure series
Population: one subject withdrawal from each group due to personal reasons
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sham Treatment: Subject will breathe air at less than 1.3 Atmospheres Absolute (ATA) in three 30 minute periods separated by 10 minutes of breathing air at less that 1.3 ATA. Hyperbaric exposures will be done up to 5 times per week with a total number of 30 exposures.
  Sham treatment
Arm/Group | Sham Treatment | Hyperbaric Oxygen 2.4 ATA
Number analyzed (Participants) | 24 | 24
units on a scale
  Baseline | 70.48 (13.05) | 74.21 (12.03)
  six weeks post hyperbaric exposure series | 78.12 (16.087) | 75.36 (15.230)

2. Primary Outcome: Posttraumatic Stress Disorder Checklist - Military Version (PCL-M) Scores
Description: The PCL-M is a self reported test in which a list of 17 problems and complaints are offered to the individual to score on a 1 to 5 scale with 1 designating "not at all", 2= "a little bit", 3= "moderately", 4= "quite a bit" and 5 designating "extremely". A sample complaint would be "repeated, disturbing dreams of a stressful military experience". Hence there is a possible total score range from 17 to 85. For military members, a score of 50 or above is indicative of PTSD. A change from baseline of 5-9 represents a reliable change and change of 10 or greater is a significant change.
Time Frame: baseline compared to the change at post hyperbaric exposures (30) series and the six weeks post hyperbaric exposure series
Population: Per protocol. The study was a pilot.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Treatment | Hyperbaric Oxygen 2.4 ATA
Number analyzed (Participants) | 24 | 24
units on a scale
  Baseline measurement | 48.88 (12.59) | 50.38 (14.53)
  Post 30 hyperbaric exposures | -10.125 (10.759) | -8.875 (8.789)
  6 Week Follow-up | -8.292 (10.960) | -8.625 (10.761)
Statistical Analysis 1: Comparison: Sham Treatment vs Hyperbaric Oxygen 2.4 ATA; ANCOVA, baseline measurement was considered as a covariate and group (sham or 2.4 ATA), treatment (15 treatments, 30 treatments, and 6 weeks) as well as the interaction between group and treatment were considered as the independent variables; Test type: Superiority or Other; p = 0.05, ANCOVA; A repeated measures model was designed so as to incorporate the adjust for the repeated (dependent) measures within individuals over time

3. Primary Outcome: Computer Cognitive Test Scores - ImPACT Visual Memory
Description: The Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT) battery was developed at the University of Pittsburgh. It has a sensitivity of 81.9% and specificity of 89.4% in discriminating between concussion and non-concussion groups. It consists of a medical history questionnaire regarding concussions and resultant symptoms including loss of consciousness, memory loss, confusion, headache, seizure activity, emotional state, and sleep patterns. There are four subtests given and scored by computer. These include verbal and visual memory, visual motor speed, and response time. The composite scores are specifically designed to determine changes within the individual, better or worse, over time. The visual memory score demonstrates improvement as the score increases. The score range was 31.2 to 92.7.
Time Frame: Baseline and six weeks post hyperbaric exposure series
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Treatment | Hyperbaric Oxygen 2.4 ATA
Number analyzed (Participants) | 24 | 24
units on a scale
  Baseline | 56.56 (14.86) | 59.8 (12.17)
  six weeks post hyperbaric exposure series | 64.72 (15.19) | 66.8 (14.72)

4. Primary Outcome: Computer Cognitive Test Scores - ImPACT Processing Speed
Description: The Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT) battery was developed at the University of Pittsburgh. It has a sensitivity of 81.9% and specificity of 89.4% in discriminating between concussion and non-concussion groups. It consists of a medical history questionnaire regarding concussions and resultant symptoms including loss of consciousness, memory loss, confusion, headache, seizure activity, emotional state, and sleep patterns. There are four subtests given and scored by computer. These include verbal and visual memory, visual motor speed, and response time. The composite scores are specifically designed to determine changes within the individual, better or worse, over time. The Processing Speed score demonstrates improvement as the score increases. The score range was 9.7 to 52.4.
Time Frame: Baseline and six weeks post hyperbaric exposure series
Population: one subject withdrawal from each group due to personal reasons
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Treatment | Hyperbaric Oxygen 2.4 ATA
Number analyzed (Participants) | 24 | 24
units on a scale
  Baseline | 30.26 (8.50) | 29.62 (9.61)
  Six weeks post hyperbaric exposure series | 36.71 (10.47) | 33.84 (10.30)

5. Primary Outcome: Computer Cognitive Test Scores - ImPACT Reaction Time
Description: The Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT) battery was developed at the University of Pittsburgh. It has a sensitivity of 81.9% and specificity of 89.4% in discriminating between concussion and non-concussion groups. It consists of a medical history questionnaire regarding concussions and resultant symptoms including loss of consciousness, memory loss, confusion, headache, seizure activity, emotional state, and sleep patterns. There are four subtests given and scored by computer. These include verbal and visual memory, visual motor speed, and response time. The composite scores are specifically designed to determine changes within the individual, better or worse, over time. The reaction time score demonstrates improvement as the score decreases. The score range was 0.42 to 1.84.
Time Frame: Baseline and six weeks post hyperbaric exposure series
Population: one subject withdrawal from each group due to personal reasons
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Treatment | Hyperbaric Oxygen 2.4 ATA
Number analyzed (Participants) | 24 | 24
units on a scale
  Baseline | 0.739 (0.322) | 0.725 (0.199)
  Six weeks post hyperbaric exposure series | 0.677 (0.186) | 0.712 (0.266)

6. Primary Outcome: Computer Cognitive Test Scores - BrainCheckers Simple Reaction Time
Description: Braincheckers is a PDA version of the Automated Neuropsychological Assessment Metrics (ANAM) supported by the Army Medical Research and Materiel Command in 2000. It was validated against ANAM for the individual tests used. Throughput is defined as correct responses per minute of time available to respond. Higher scores indicate higher accuracy in each of the subtest. The simple reaction time range is 30 to 255.
Time Frame: Baseline and six weeks post hyperbaric exposure series
Population: One subject withdrawal from each group due to personal reasons
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Treatment | Hyperbaric Oxygen 2.4 ATA
Number analyzed (Participants) | 24 | 24
units on a scale
  Baseline | 142.21 (60.68) | 135.79 (61.48)
  Six weeks post hyperbaric exposure series | 174.96 (57.75) | 171.83 (54.66)

7. Primary Outcome: Computer Cognitive Test Scores - BrainCheckers Code Substitution
Description: Braincheckers is a PDA version of the Automated Neuropsychological Assessment Metrics (ANAM) supported by the Army Medical Research and Materiel Command in 2000. It was validated against ANAM for the individual tests used. Throughput is defined as correct responses per minute of time available to respond. Higher scores indicate higher accuracy in each of the subtest. The range is 9 to 66. The scores in this section represent results of the code substitution subtest.
Time Frame: Baseline and six weeks post hyperbaric exposure series
Population: One subject withdrawal from each group due to personal reasons
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Treatment | Hyperbaric Oxygen 2.4 ATA
Number analyzed (Participants) | 24 | 24
units on a scale
  Baeline | 39.20 (12.08) | 37.42 (13.74)
  Post hyperbaric exposure 6 week follow up throughp | 43.39 (13.56) | 40.71 (12.10)

8. Primary Outcome: Computer Cognitive Test Scores - BrainCheckers Procedural Reaction Time
Description: Braincheckers is a PDA version of the Automated Neuropsychological Assessment Metrics (ANAM) supported by the Army Medical Research and Materiel Command in 2000. It was validated against ANAM for the individual tests used. Throughput is defined as correct responses per minute of time available to respond. Higher scores indicate higher accuracy in each of the subtest. The range is 25 to 118. The scores in this section represent results of the procedural reaction time.
Time Frame: Baseline and six weeks post hyperbaric exposure series
Population: One subject withdrawal from each group due to personal reasons
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Treatment | Hyperbaric Oxygen 2.4 ATA
Number analyzed (Participants) | 24 | 24
units on a scale
  Baseline | 81.63 (20.82) | 81.17 (21.66)
  Post hyperbaric exposure 6 week follow up throughp | 85.78 (23.16) | 86.78 (16.63)

9. Primary Outcome: Computer Cognitive Test Scores - BrainCheckers Go-NoGo Reaction Time
Description: Braincheckers is a PDA version of the Automated Neuropsychological Assessment Metrics (ANAM) supported by the Army Medical Research and Materiel Command in 2000. It was validated against ANAM for the individual tests used. Throughput is defined as correct responses per minute of time available to respond. Higher scores indicate higher accuracy in each of the subtest. The range is 41 to 174. The scores in this section represent results of the Go-NoGo reaction time subtest.
Time Frame: Baseline and six weeks post hyperbaric exposure series
Population: One subject withdrawal from each group due to personal reasons
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Treatment | Hyperbaric Oxygen 2.4 ATA
Number analyzed (Participants) | 24 | 24
units on a scale
  Baseline | 119.67 (31.03) | 116.52 (23.33)
  Post hyperbaric exposure 6 week follow up throughp | 131.70 (31.43) | 129.17 (25.67)

10. Primary Outcome: Computer Cognitive Test Scores - BrainCheckers Matching To Sample
Description: BrainCheckers is a PDA version of the Automated Neuropsychological Assessment Metrics (ANAM) supported by the Army Medical Research and Materiel Command in 2000. It was validated against ANAM for the individual tests used. Throughput is defined as correct responses per minute of time available to respond. Higher scores indicate accuracy in each of the subtest. The range is 6 to 50. The scores in this section represent results of the matching to sample subtest.
Time Frame: Baseline and six weeks post hyperbaric exposure series
Population: One subject withdrawal from each group due to personal reasons
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Treatment | Hyperbaric Oxygen 2.4 ATA
Number analyzed (Participants) | 24 | 24
units on a scale
  Baseline | 20.00 (10.70) | 23.71 (11.86)
  Post hyperbaric exposure 6 week follow up throughp | 28.22 (10.63) | 24.42 (8.08)

11. Primary Outcome: Computer Cognitive Test Scores - BrainCheckers Code Sub Recall
Description: BrainCheckers is a PDA version of the Automated Neuropsychological Assessment Metrics (ANAM) supported by the Army Medical Research and Materiel Command in 2000. It was validated against ANAM for the individual tests used. Throughput is defined as correct responses per minute of time available to respond. Higher scores indicate accuracy in each of the subtest. The range is 6 to 135. The scores in this section represent results of the code sub recall subtest.
Time Frame: Baseline and six weeks post hyperbaric exposure series
Population: One subject withdrawal from each group due to personal reasons
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham Treatment | Hyperbaric Oxygen 2.4 ATA
Number analyzed (Participants) | 24 | 24
units on a scale
  Baseline | 29.88 (16.63) | 36.38 (19.77)
  Post hyperbaric exposure 6 week follow up throughp | 47.57 (24.02) | 44.08 (12.07)

12. Secondary Outcome: Functional MRI
Time Frame: six weeks post hyperbaric exposure series
Reporting Status: Not Posted

13. Secondary Outcome: Stem Cells: CD_34
Description: A non-parametric regression 14 using the Theil estimator was fit to the observed data in order to demonstrate general trends for relations between measures of cognitive functioning and increased stem cells.
Time Frame: six weeks post hyperbaric exposure series
Reporting Status: Not Posted

14. Post Hoc Outcome: PCL-M Relative Risk of Improvement of 2.4 ATA Exposures vs. Sham, All Participants With Only One Concussive Event
Description: The purpose of a pilot study is to identify potential subgroups who may respond to treatment. The various composite scores were ranked and separated by subject and within groups for those who improved and those who did not. This allowed the application relative risk analysis using MedCalc (http://www.medcalc.org) to identify potential subgroups. Relative Risk of Improvement (RROI) was calculated against the concussion history items. Main categories were the number of concussive events, whether the subject had multiple non-concussive events or not, if there were two concussive events within a 48 hour period, the time expired from the last concussion to consent, the etiology of the event, and loss of consciousness. A concussive event was defined as one immediately followed with symptoms. This outcome measure analyzed PCL-M score decreases of 10 or more (significantly improved) in the individuals who experienced only one concussive event.
Time Frame: Baseline values compared to 30 post hyperbaric exposure or 6 week follow-up
Population: Participants with significant improvement (PCL-M composite scores demonstrating a decrease by 10 or greater) or participants not meeting this criterion.
Measure: Number; unit: participants
Groups:
- Sham Treatment Improved: Subjects breathed air at less than 1.3 Atmospheres Absolute (ATA) in three 30 minute periods separated by 10 minutes of breathing air at less that 1.3 ATA. See previous description for details.
  PCL-M composite scores demonstrated a significant (decrease by10 or greater)improvement or a reliable (decrease by 5 or greater) from baseline at 30 post hyperbaric exposure or 6 week follow-up.
- Sham Treatment Not Improved: Subjects breathed air at less than 1.3 Atmospheres Absolute (ATA) in three 30 minute periods separated by 10 minutes of breathing air at less that 1.3 ATA. See previous description for details.
  PCL-M composite scores demonstrated a decrease of 4 or less from baseline at 30 post hyperbaric exposure or 6 week follow-up.
- Hyperbaric Oxygen 2.4 ATA Improved: Subject breathed 100% oxygen at 2.4 Atmospheres Absolute (ATA) in three 30 minute periods separated by 10 minutes of breathing air at 2.4 ATA. See previous description for details.
  PCL-M composite scores demonstrated a significant (decrease by10 or greater)improvement or a reliable (decrease by 5 or greater) from baseline at 30 post hyperbaric exposure or 6 week follow-up.
- Hyperbaric Oxygen 2.4 ATA Not Improved: Subject breathed 100% oxygen at 2.4 Atmospheres Absolute (ATA) in three 30 minute periods separated by 10 minutes of breathing air at 2.4 ATA. See previous description for details.
  PCL-M composite scores demonstrated a decrease of 4 or less from baseline at 30 post hyperbaric exposure or 6 week follow-up.
Arm/Group | Sham Treatment Improved | Sham Treatment Not Improved | Hyperbaric Oxygen 2.4 ATA Improved | Hyperbaric Oxygen 2.4 ATA Not Improved
Number analyzed (Participants) | 15 | 9 | 13 | 11
participants | 4 | 2 | 4 | 7
Statistical Analysis 1: Comparison: Sham Treatment Improved vs Sham Treatment Not Improved vs Hyperbaric Oxygen 2.4 ATA Improved vs Hyperbaric Oxygen 2.4 ATA Not Improved; Relative Risk of Improvement in 2.4 ATA group vs. Sham in subjects with one significant event (blast or impact resulting in concussion symptoms) per Concussion History. PCL-M with significant improvement defined as a score decrease 10 or more; Test type: Superiority or Other; Risk Ratio (RR) = 0.5455

15. Post Hoc Outcome: PCL-M Relative Risk of Improvement of 2.4 ATA Exposures vs. Sham, All Participants With Two Concussive Events
Description: The purpose of a pilot study is to identify potential subgroups who may respond to treatment. The various composite scores were ranked and separated by subject and within groups for those who improved and those who did not. This allowed the application relative risk analysis using MedCalc (http://www.medcalc.org) to identify potential subgroups. Relative Risk of Improvement (RROI) was calculated against the concussion history items. Main categories were the number of concussive events, whether the subject had multiple non-concussive events or not, if there were two concussive events within a 48 hour period, the time expired from the last concussion to consent, the etiology of the event, and loss of consciousness. A concussive event was defined as one immediately followed with symptoms. This outcome measure analyzed PCL-M score decreases of 10 or more (significantly improved) in individuals who experienced two concussive events.
Time Frame: Baseline values compared to 30 post hyperbaric exposure or 6 week follow-up
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Sham Treatment Improved | Sham Treatment Not Improved | Hyperbaric Oxygen 2.4 ATA Improved | Hyperbaric Oxygen 2.4 ATA Not Improved
Number analyzed (Participants) | 15 | 9 | 13 | 11
participants | 6 | 5 | 3 | 2
Statistical Analysis 1: Comparison: Sham Treatment Improved vs Sham Treatment Not Improved vs Hyperbaric Oxygen 2.4 ATA Improved vs Hyperbaric Oxygen 2.4 ATA Not Improved; Relative Risk of Improvement in 2.4 ATA group vs. Sham in subjects with two significant events (blast or impact resulting in concussion symptoms) per Concussion History. PCL-M with significant improvement defined as a score decrease 10 or more; Test type: Superiority or Other; Risk Ratio (RR) = 1.10

16. Post Hoc Outcome: PCL-M Relative Risk of Improvement of 2.4 ATA Exposures vs. Sham, All Participants With Three Concussive Events
Description: The purpose of a pilot study is to identify potential subgroups who may respond to treatment. The various composite scores were ranked and separated by subject and within groups for those who improved and those who did not. This allowed the application relative risk analysis using MedCalc (http://www.medcalc.org) to identify potential subgroups. Relative Risk of Improvement (RROI) was calculated against the concussion history items. Main categories were the number of concussive events, whether the subject had multiple non-concussive events or not, if there were two concussive events within a 48 hour period, the time expired from the last concussion to consent, the etiology of the event, and loss of consciousness. A concussive event was defined as one immediately followed with symptoms. This outcome measure analyzed PCL-M score decreases of 10 or more (significantly improved) in individuals who experienced three concussive events.
Time Frame: Baseline values compared to 30 post hyperbaric exposure or 6 week follow-up
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Sham Treatment Improved | Sham Treatment Not Improved | Hyperbaric Oxygen 2.4 ATA Improved | Hyperbaric Oxygen 2.4 ATA Not Improved
Number analyzed (Participants) | 15 | 9 | 13 | 11
participants | 3 | 2 | 4 | 2
Statistical Analysis 1: Comparison: Sham Treatment Improved vs Sham Treatment Not Improved vs Hyperbaric Oxygen 2.4 ATA Improved vs Hyperbaric Oxygen 2.4 ATA Not Improved; Relative Risk of Improvement in 2.4 ATA group vs. Sham in subjects with three significant events (blast or impact resulting in concussion symptoms) per Concussion History. PCL-M with significant improvement defined as a score decrease 10 or more; Test type: Superiority or Other; Risk Ratio (RR) = 1.1111

17. Post Hoc Outcome: PCL-M Relative Risk of Improvement of 2.4 ATA Exposures vs. Sham, All Participants With Four or More Concussive Events
Description: The purpose of a pilot study is to identify potential subgroups who may respond to treatment. The various composite scores were ranked and separated by subject and within groups for those who improved and those who did not. This allowed the application relative risk analysis using MedCalc (http://www.medcalc.org) to identify potential subgroups. Relative Risk of Improvement (RROI) was calculated against the concussion history items. Main categories were the number of concussive events, whether the subject had multiple non-concussive events or not, if there were two concussive events within a 48 hour period, the time expired from the last concussion to consent, the etiology of the event, and loss of consciousness. A concussive event was defined as one immediately followed with symptoms. This outcome measure analyzed PCL-M score decreases of 10 or more (significantly improved) in individuals who experienced four or more concussive events.
Time Frame: Baseline values compared to 30 post hyperbaric exposure or 6 week follow-up
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Sham Treatment Improved | Sham Treatment Not Improved | Hyperbaric Oxygen 2.4 ATA Improved | Hyperbaric Oxygen 2.4 ATA Not Improved
Number analyzed (Participants) | 15 | 9 | 13 | 11
participants | 2 | 0 | 2 | 0
Statistical Analysis 1: Comparison: Sham Treatment Improved vs Sham Treatment Not Improved vs Hyperbaric Oxygen 2.4 ATA Improved vs Hyperbaric Oxygen 2.4 ATA Not Improved; Relative Risk of Improvement in 2.4 ATA group vs. Sham in subjects with four or more significant events (blast or impact resulting in concussion symptoms) per Concussion History. PCL-M with significant improvement defined as a score decrease 10 or more; Test type: Superiority or Other; Risk Ratio (RR) = 1.0

18. Post Hoc Outcome: PCL-M Relative Risk of Improvement of 2.4 ATA Exposures vs. Sham, All Participants With Multiple Non-concussive Blast and/or Impact Exposures.
Description: The purpose of a pilot study is to identify potential subgroups who may respond to treatment. The various composite scores were ranked and separated by subject and within groups for those who improved and those who did not. This allowed the application relative risk analysis using MedCalc (http://www.medcalc.org) to identify potential subgroups. Relative Risk of Improvement (RROI) was calculated for the number of concussive events, whether the subject had multiple non-concussive events or not, if there were two concussive events within a 48 hour period, the time expired from the last concussion to consent, the etiology of the event, and loss of consciousness. Many subjects had multiple blast and/or impact events without a concussion (asymptomatic), but had a flight or flight (danger response) experience. This outcome measure analyzed PCL-M score decreases of 10 or more (significantly improved) in individuals who experienced multiple non-concussive blast and/or impact events.
Time Frame: Baseline values compared to 30 post hyperbaric exposure or 6 week follow-up
Population: Participants with significant improvement (PCL-M composite scores demonstrating a decrease by 10 or greater) or participants not meeting this criterion who had multiple blast and/or impact event that did not result in a concussion (asymptomatic), but had a flight or flight (danger response) experience.
Measure: Number; unit: participants
Groups:
- Sham Treatment Improved: Subjects breathed air at less than 1.3 Atmospheres Absolute (ATA) in three 30 minute periods separated by 10 minutes of breathing air at less that 1.3 ATA. See previous description for details.
  PCL-M composite scores demonstrated a significant (decrease by10 or greater)improvement from baseline at 30 post hyperbaric exposure or 6 week follow-up.
- Sham Treatment Not Improved: Subjects breathed air at less than 1.3 Atmospheres Absolute (ATA) in three 30 minute periods separated by 10 minutes of breathing air at less that 1.3 ATA. See previous description for details.
  PCL-M composite scores demonstrated a significant (decrease by 9 or less)improvement from baseline at 30 post hyperbaric exposure or 6 week follow-up.
- Hyperbaric Oxygen 2.4 ATA Improved: Subject breathed 100% oxygen at 2.4 Atmospheres Absolute (ATA) in three 30 minute periods separated by 10 minutes of breathing air at 2.4 ATA. See previous description for details.
  PCL-M composite scores demonstrated a significant (decrease by10 or greater)improvement from baseline at 30 post hyperbaric exposure or 6 week follow-up.
- Hyperbaric Oxygen 2.4 ATA Not Improved: Subject breathed 100% oxygen at 2.4 Atmospheres Absolute (ATA) in three 30 minute periods separated by 10 minutes of breathing air at 2.4 ATA. See previous description for details.
  PCL-M composite scores demonstrated a significant (decrease by 9 or less)improvement from baseline at 30 post hyperbaric exposure or 6 week follow-up.
Arm/Group | Sham Treatment Improved | Sham Treatment Not Improved | Hyperbaric Oxygen 2.4 ATA Improved | Hyperbaric Oxygen 2.4 ATA Not Improved
Number analyzed (Participants) | 17 | 7 | 7 | 17
participants | 11 | 5 | 2 | 9

19. Post Hoc Outcome: PCL-M Relative Risk of Improvement of 2.4 ATA Exposures vs. Sham, Measuring Time to Consent From the Last Concussion in Subjects With Multiple Concussions.
Description: The purpose of a pilot study is to identify potential subgroups who may respond to treatment. The various composite scores were ranked and separated by subject and within groups for those who improved and those who did not. This allowed the application relative risk analysis using MedCalc (http://www.medcalc.org) to identify potential subgroups. Relative Risk of Improvement (RROI) was calculated for the number of concussive events, whether the subject had multiple non-concussive events or not, if there were two concussive events within a 48 hour period, the time expired from the last concussion to consent, the etiology of the event, and loss of consciousness. This outcome measure analyzed PCL-M score decreases of 10 or more (significantly improved) with consent within one year from the last concussion in subjects who had multiple concussions.
Time Frame: Baseline values compared to 30 post hyperbaric exposure or 6 week follow-up
Measure: Number; unit: participants
Groups:
- Sham Treatment Not Improved: Subjects breathed air at less than 1.3 Atmospheres Absolute (ATA) in three 30 minute periods separated by 10 minutes of breathing air at less that 1.3 ATA. See previous description for details.
  PCL-M composite scores demonstrated a decrease of 9 or less from baseline at 30 post hyperbaric exposure or 6 week follow-up.
- Hyperbaric Oxygen 2.4 ATA Not Improved: Subject breathed 100% oxygen at 2.4 Atmospheres Absolute (ATA) in three 30 minute periods separated by 10 minutes of breathing air at 2.4 ATA. See previous description for details.
  PCL-M composite scores demonstrated a decrease of 9 or less from baseline at 30 post hyperbaric exposure or 6 week follow-up.
Arm/Group | Sham Treatment Improved | Sham Treatment Not Improved | Hyperbaric Oxygen 2.4 ATA Improved | Hyperbaric Oxygen 2.4 ATA Not Improved
Number analyzed (Participants) | 17 | 7 | 17 | 7
participants | 1 | 3 | 3 | 2

ADVERSE EVENTS:
Arm/Group | Sham Treatment | Hyperbaric Oxygen 2.4 ATA
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 4/25 | 10/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Treatment (N=25) | Hyperbaric Oxygen 2.4 ATA (N=25)
Ear block (Ear and labyrinth disorders) | 4 (8) | 10 (44) — Ear blocks - subject unable to equalize middle ear pressure during descent requiring the pressurization to be stopped. Blocks/exposures rate - sham: 0.01; treatment: 0.06. Subject post exams with TEED 2 or less using 0-5 scale.

LIMITATIONS AND CAVEATS:
Caveats: Analysis used both repeated measures of analysis of covariance (ANCOVA) and repeated measures analysis of variance (RMANOVA). Due to the results, analysis is currently identifying potential subgroups which may demonstrate significance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes